CLINICAL TRIAL: NCT01051414
Title: A Phase 2a Study of BMS-790052 and BMS-650032 in Combination Therapy With Japanese Subjects With Genotype 1 Chronic Hepatitis C (HCV) Virus Infection
Brief Title: An Anti-viral Combination Study With Japanese Hepatitis C Infection (HCV) Subject
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI447-017
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-790052 + BMS-650032 (Experimental)
  Interventions: Drug: BMS-790052; Drug: BMS-650032

INTERVENTIONS:
Drug: BMS-790052 — Tablets, Oral, 60 mg, daily, 24 weeks
Drug: BMS-650032 — Tablets, Oral, 1200 mg, daily, 24 weeks

SUMMARY:
To assess the efficacy and safety profile of co-administration of BMS-790052 and BMS-650032 for 24 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects chronically infected with HCV Genotype 1
* HCV RNA viral load of ≥ 10*5* IU/mL (100,000 IU/mL) at screening

Exclusion Criteria:

* Subjects with evidence of liver cirrhosis
* Evidence of HCC
* Co-infection with hepatitis B virus, HIV

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Part 1: To assess safety and tolerability based on 4 weeks safety data, as measured by related serious adverse events (SAEs) and discontinuations due to related AEs | Week 4
Part 2: To determine the proportion of subjects who achieve SVR12 (i.e., HCV RNA < 15 IU/mL at follow-up Week 12) | Post-treatment Week 12

SECONDARY OUTCOMES:
The safety of co-administration of BMS-790052 + BMS-650032 as measured by the frequency of SAEs, discontinuations due to AEs, and Grade 3 - 4 laboratory abnormalities | Weeks 4, 12, end of treatment and post-treatment Week 24
The proportion of subjects who achieve RVR (defined as HCV RNA < 15 IU/mL | Week 4
The proportion of subjects with extended rapid virologic response (eRVR), defined as HCV RNA < 15 IU/mL | at both Weeks 4 and 12
The proportion of subjects who achieve SVR24 (defined as HCV RNA < 15 IU/mL | at follow-up Week 24
Resistant variants associated with clinical failure | Weeks 4, 12, end of treatment and post-treatment Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Japan (4):
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kawasaki-Shi, Kanagawa
  - Local Institution, Minato-Ku, Tokyo

REFERENCES:
- [Derived] Kao JH, Jensen DM, Manns MP, Jacobson I, Kumada H, Toyota J, Heo J, Yoffe B, Sievert W, Bessone F, Peng CY, Roberts SK, Lee YJ, Bhore R, Mendez P, Hughes E, Noviello S. Daclatasvir plus asunaprevir for HCV genotype 1b infection in patients with or without compensated cirrhosis: a pooled analysis. Liver Int. 2016 Jul;36(7):954-62. doi: 10.1111/liv.13049. Epub 2016 Jan 24. PMID 26683763
- [Derived] Suzuki Y, Ikeda K, Suzuki F, Toyota J, Karino Y, Chayama K, Kawakami Y, Ishikawa H, Watanabe H, Hu W, Eley T, McPhee F, Hughes E, Kumada H. Dual oral therapy with daclatasvir and asunaprevir for patients with HCV genotype 1b infection and limited treatment options. J Hepatol. 2013 Apr;58(4):655-62. doi: 10.1016/j.jhep.2012.09.037. Epub 2012 Nov 23. PMID 23183526
- [Derived] Karino Y, Toyota J, Ikeda K, Suzuki F, Chayama K, Kawakami Y, Ishikawa H, Watanabe H, Hernandez D, Yu F, McPhee F, Kumada H. Characterization of virologic escape in hepatitis C virus genotype 1b patients treated with the direct-acting antivirals daclatasvir and asunaprevir. J Hepatol. 2013 Apr;58(4):646-54. doi: 10.1016/j.jhep.2012.11.012. Epub 2012 Nov 22. PMID 23178977
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx